CLINICAL TRIAL: NCT06615609
Title: "Smart Family Doctor" Assisted Comprehensive Management of Secondary Prevention Among Post Coronary Artery Bypass Graft Patients or Post Percutaneous Coronary Intervention Patients
Acronym: SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Xin Yuan, Professor, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FW-YX-001
Record Dates: First submitted 2024-09-21; First posted 2024-09-26 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Post Coronary Artery Bypass Grafting; Hypertension; Diabetes Mellitus; Hyperlipidemia; Post PCI
Keywords: smartphone; AI-assisted; CABG management; metabolic management; Smart family doctor
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: The intervention in this study is the implementation of the 'Smart family doctor' system, a digital health management tool designed to support secondary prevention in post-CABG patients or post-PCI patients. This system leverages knowledge from coronary artery disease (CAD) secondary prevention guidelines, expert consensus, and a knowledge base addressing common post-CABG issues. It is powered by a large-scale, medical knowledge-enhanced conversational model, enabling personalized interactions with patients to guide their recovery and lifestyle management following surgery.
Masking Description: Data manager and statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Smart family doctor" assisted management plus health managers (Experimental): "Smart family doctor", an AI-assisted applications with personalized interactions and 3-hour health management guidance from a health manager once a week.
  Interventions: Behavioral: Smart family doctor; Behavioral: Health manager
- Usual care: health managers (Placebo Comparator): 3-hour health management guidance from a health manager once a week.
  Interventions: Behavioral: Health manager

INTERVENTIONS:
Behavioral: Smart family doctor — Based on health managers, participants were additionally provided "Smart family doctor", which is an AI-assisted applications with personalized interactions. The content includes, but is not limited to: (1) General educational content, covering basic health knowledge on diseases, risk factors, and treatment methods; (2) Targeted health information, such as more specific guidance on blood pressure and blood sugar control, medication adherence, exercise, and smoking cessation; (3) Personalized disease management guidance, providing tailored reminders for patients regarding medication, diet, exercise, and medical visits. Patients can also directly report their latest self-measured blood pressure, blood lipid, blood sugar levels, and medication adherence to receive treatment and medication guidance from the 'Smart family doctor'.
  Arms: "Smart family doctor" assisted management plus health managers
Behavioral: Health manager — Participants will received 3-hour health management guidance from a health manager once a week, including guidance on healthy lifestyle, medication treatment, and rehabilitation advice. The research team will provide participants with one smart band, requiring them to wear the band daily to collect health data during the 6-month study period.

SUMMARY:
This study aims to evaluate the effect of an AI-assisted "Smart family doctor" digital health management tool on improving the control rates of hypertension, diabetes, and dyslipidemia in post-CABG (coronary artery bypass grafting) patients or post-PCI (percutaneous coronary intervention) patients. A randomized controlled trial design will be used, involving approximately 5-10 hospitals and 536 participants. Eligible participants are adults aged 18 or older, post-CABG or post-PCI patients with hypertension, diabetes, and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* History of CABG surgery or PCI with history of hypertension, diabetes, and dyslipidemia.
* At least one of the following criteria is meet:
* Systolic blood pressure no less than 130 mmHg or diastolic blood pressure no less than 80 mmHg
* HbA1c no less than 7%
* LDL-C no less than 1.4 mmol/L
* Use of a smartphone.
* Signed informed consent.

Exclusion Criteria:

* History of heart failure or severe arrhythmias.
* Presence of other severe underlying conditions such as cancer or liver and kidney insufficiency.
* Pregnancy, lactation, or plans for pregnancy within the next year.
* Cognitive, communication impairments, or limitations in daily activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
The control rates of hypertension, diabetes and hyperlipidemia | 6-month
  All cretria are meet:
  1. Systolic blood pressure less than 130 mmHg and diastolic blood pressure less than 80 mmHg.
  2. HbA1c less than 7%.
  3. LDL-C less than 1.4 mmol/L.

SECONDARY OUTCOMES:
Blood Pressure Control Rate | 6-month
  The proportion of patients with systolic blood pressure less than 130 mmHg and diastolic blood pressure less than 80 mmHg.
Smoking Rate | 6-month
  The proportion of patients who have smoked within the past month.
Total cholesterol | 6-month
  Total cholesterol analyzed at central lab.
LDL-C | 6-month
  LDL-C analyzed at central lab.
HDL-C | 6-month
  HDL-C analyzed at central lab.
Triglycerides | 6-month
  Triglycerides analyzed at central lab.
Small dense LDL-C | 6-month
  Small dense LDL-C analyzed at central lab.
Lipoprotein (a) | 6-month
  Lipoprotein (a) analyzed at central lab.
Fasting blood glucose | 6-month
  Fasting blood glucose analyzed at central lab.
HbA1c | 6-month
  HbA1c levels analyzed at central lab.
Physical Activity Level | 6-month
  Assessed using the International Physical Activity Questionnaire (IPAQ) and decribed as total MET of walking, moderate, or high intensity physical activity.
Quality of life using the Short Form Health Survey (SF-12v2) | 6-month
  Quality of life using the Short Form Health Survey (SF-12v2). The higher score indicated the better quality of life.
Coronary artery disease-related quality of life | 6-month
  Coronary artery disease-related quality of life assessed with the Seattle Angina Questionnaire (SAQ). The higher score indicated the better coronary artery disease-related quality of life.
Psychological status | 6-month
  Psychological status evaluated using the 9-item Patient Health Questionnaire (PHQ-9). The higher score indicated the worse psychological status
Cognitive function | 6-month
  Cognitive function assessed with the Mini-Cog test. The higher score indicated the better conginition.

OTHER OUTCOMES:
Major adverse cardiovascular events (MACE) | 6-month
  The composite endpoint of cardiovascular death, myocardial infarction, stroke, or hospitalization due to cardiovascular disease.
C-reactive protein | 6-month
  C-reactive protein (CRP) analyzed at central lab.
interleukin-6 | 6-month
  Interleukin-6 (IL-6) is analyzed at central lab.
Interleukin-10 | 6-month
  Interleukin-10 (IL-10) is analyzed at central lab.
Interleukin-1β (IL-1β) | 6-month
  Interleukin-1β (IL-1β) is analyzed at central lab.
tumor necrosis factor-α (TNF-α) | 6-month
  Tumor necrosis factor-α (TNF-α) is analyzed at central lab.
prostaglandin | 6-month
  prostaglandin (PG) is analyzed at central lab.
Intercellular adhesion molecule-1 | 6-month
  Intercellular adhesion molecule-1 (ICAM-1) is analysed at central lab.
Von Willebrand factor | 6-month
  Von Willebrand factor (vWF) is analyzed at central lab.
Urinary albumin-to-creatinine ratio | 6-month
  Urinary albumin-to-creatinine ratio is calculated as urine albumin divided by urine creatinine.
Urinary sodium excretion rate | 6-month
  Urinary sodium excretion rate is analyzed at central lab.
BMI | 6-month
  Body mass index (BMI) is calculated as weights (kg) divided by the square of heights (meters).
Waist circumference | 6-month
  Waist circumference is measured at local site.
Cost-effectiveness analysis | 6-month
  The incremental cost-effectiveness ratio (ICER): the additional cost per patient achieving target control of hypertension, dyslipidemia, or diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Yuan, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Xinjiang's First Affiliated Hospital of medical university, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data that support the findings of this study are available from the corresponding author, upon reasonable request, only for authorized research. Their use is subjected to an agreement with the promotor (Fuwai Hospital) and the principal investigator (Dr Xin Yuan) of the SMART study. Pseudonymised data that support the findings of this study are available from the promotor (Fuwai Hospital) upon reasonable request, subject to a specific agreement with the promotor (involving the principal investigator) and subject to regulatory proceedings due to data protection applicable laws. Access conditions are to be determined depending on the nature of the request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the end of the study
Access Criteria: Anonymized data that support the findings of this study are available from the corresponding author, upon reasonable request, only for authorized research. Their use is subjected to an agreement with the promotor (Fuwai Hospital) and the principal investigator (Dr Xin Yuan) of the SMART study. Pseudonymised data that support the findings of this study are available from the promotor (Fuwai Hospital) upon reasonable request, subject to a specific agreement with the promotor (involving the principal investigator) and subject to regulatory proceedings due to data protection applicable laws. Access conditions are to be determined depending on the nature of the request.

REFERENCES:
- [Derived] Lei L, Li J, Zhang L, Yuan X, Diao X, Qi L, Wang Y, Du W, Zhao W, Hu S. Design and rationale of the artificial intelligent dialogue System assisted comprehensive Management of secondary prevention Among post coronary aRtery bypass graft patienTs (SMART): protocol for a randomised controlled trial for postcoronary artery bypass grafting management. BMJ Open. 2025 Nov 11;15(11):e106447. doi: 10.1136/bmjopen-2025-106447. PMID 41218945